CLINICAL TRIAL: NCT04084041
Title: Efficacy of the Simeox Airway Clearance Technology in the Treatment of Children With Clinically Stable Cystic Fibrosis- Cross-over Study With Randomization
Brief Title: Efficacy of Simeox Airway Clearance Therapy in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Assist (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HOMECARE_CF
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis in Children; Airway Clearance Impairment
Keywords: Airway clearance technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device (Experimental): Device group
  Interventions: Device: Simeox; Other: CCPT
- Conventional chest physiotherapy (Active Comparator): Control group
  Interventions: Device: Simeox; Other: CCPT

INTERVENTIONS:
Device: Simeox — Airway clearance device
Other: CCPT — Conventional chest physiotherapy

SUMMARY:
Chest physiotherapy plays a crucial role in treatment of lung disease in cystic fibrosis (CF). New airway clearance techniques (ACTs) adapted to individual needs are still being sought to achieve the best effect of airway clearance. The primary aim of this study is to assess the efficacy of a new ACT (Simeox) on pulmonary function in children with CF. 40 CF patients with stable respiratory function will be randomized 1:1 to Simeox or conventional chest physiotherapy (CCPT) therapy (control group) and treated at home during 1 month. After a short washout period, patients will be treated at home onto the alternative treatment for 1 month (crossover design). Lung function, quality of life, pulmonary exacerbation and safety will be evaluated at 1 month for each therapy period.

ELIGIBILITY:
Inclusion Criteria:

* Subject and his or her legally appointed and authorized representative will agree for treatment with Simeox technology
* willing and able to cooperate and learn new technic of drainage.
* age 8-18 years, on the date of admission to hospital.
* confirmed diagnosis of CF as determined by the investigator.
* able to perform pulmonary tests

Exclusion Criteria:

History of any illness or any clinical condition that, in the opinion of the investigator, might confound the cooperation or the results of the study or pose an additional risk to the subject in using study technology. This includes, but is not limited to, the following:

* contraindications to bronchial chest physiotherapy
* hemoptysis
* pneumothorax
* heart disease
* recent chest surgery
* recent chest injury
* history of lung transplantation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Change in total lung resistance | 1 month
  Evolution of R5hz - Impulse Oscillometry (IOS) from baseline

SECONDARY OUTCOMES:
Change in central lung resistance | 1 month
  Evolution of R20hz - Impulse Oscillometry (IOS) from baseline
Change in peripheral lung resistance | 1 month
  Evolution of R5-20hz - Impulse Oscillometry (IOS) from baseline
Change in total lung reactance | 1 month
  Evolution of X5hz -Impulse Oscillometry (IOS) from baseline
Change in area of reactance (AX) | 1 month
  Evolution of AX -Impulse Oscillometry (IOS) from baseline
Change in total score of Cystic Fibrosis Questionnaire-Revised (CFQ-R) | 1 month
  Evolution of CFQ-R total score (0-100) from baseline
Change in respiratory domain score of Cystic Fibrosis Questionnaire Revised (CFQ-R) questionnaire | 1 month
  Evolution of respiratory score (0-100) of CFQ-R from baseline
Change in Forced Expiratory Volume in 1 second (FEV1) | 1 month
  Evolution of FEV1 (spirometry) from baseline
Change in Forced Vital Capacity (FVC) | 1 month
  Evolution of FVC (spirometry) from baseline
Change in Residual Volume (RV) | 1 month
  Evolution of RV (body plethysmography) from baseline
Change in Maximal Expiratory Flow (MEF) at 25, 50 and 75% of expired volume | 1 month
  Evolution of MEF 25, 50 and 75 (spirometry) from baseline
Change in Mean Mid Expiratory Flow (MMEF) | 1 month
  Evolution of MMEF (spirometry) from baseline
Change in lung clearance index (LCI) | 1 month
  Evolution of LCI with Nitrogen multiple breath washout (N2MBW) tests from baseline
Pulmonary exacerbation | 1 month
  Rate of pulmonary exacerbation
Adverse events | 1 month
  Rate of adverse events related or not related to intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Sands, MD, PhD, Principal Investigator — IMiD
Locations (1):
- IMiD, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sands D, Walicka-Serzysko K, Milczewska J, Postek M, Jeneralska N, Cichocka A, Siedlecka E, Borawska-Kowalczyk U, Morin L. Efficacy of the Simeox(R) Airway Clearance Technology in the Homecare Treatment of Children with Clinically Stable Cystic Fibrosis: A Randomized Controlled Trial. Children (Basel). 2023 Jan 23;10(2):204. doi: 10.3390/children10020204. PMID 36832333